CLINICAL TRIAL: NCT07330115
Title: Combination of Kinesio Tape and Poprioceptive Neck Exercises on Proprioception in Patients With Cervical Radiculopathy
Brief Title: Combination of Kinesio Tape and Proprioceptive Neck Exercises on Proprioception in Patients With Cervical Radiculopathy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fadia Ahmed Fawzy (Other)
Responsible Party: Sponsor-Investigator, Fadia Ahmed Fawzy, Principal investigator, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KT and DCT on CR
Record Dates: First submitted 2025-12-17; First posted 2026-01-09 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Cervical Radiculopathy; Proprioception
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned into three parallel groups. The first group will receive proprioceptive neck exercises only, the second group will receive kinesio taping only, and the third group will receive a combination of both interventions. All groups will receive their assigned intervention throughout the study period.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- proprioceptive neck exercises group (Active Comparator): Proprioceptive neck exercises The patient will sit on a swivel chair with a backrest in front of a wall at a distance of 90 cm. A laser pointer will be fixed to the highest point of the patient's head, so the laser light will be projected on a target hanging on the wall . Then active cervical movements will be performed.
  Interventions: Other: proprioceptive neck exercises
- KT group (Active Comparator): Group B will receive KT.
  Interventions: Other: Kinesiotaping
- KT and proprioceptive neck exercises (Active Comparator): Group C will receive both (proprioceptive neck exercercises and KT)
  Interventions: Other: proprioceptive neck exercises; Other: Kinesiotaping

INTERVENTIONS:
Other: proprioceptive neck exercises — Proprioceptive craniocervical exercises The patient will sit on a swivel chair with a backrest in front of a wall at a distance of 90 cm. A laser pointer will be fixed to the highest point of the patient's head, so the laser light will be projected on a target hanging on the wall (Espí-López et al., 2020). Then active cervical movements will be performed.
  Arms: KT and proprioceptive neck exercises; proprioceptive neck exercises group
Other: Kinesiotaping — For kinesio tape application, a method of brachial plexus application will be chosen .
  Arms: KT and proprioceptive neck exercises; KT group

SUMMARY:
This study is conducted to investigate:

1. The efficiency of combination of KT and proprioceptive exercises on neck proprioception in patients with CR.
2. The efficiency of combination of KT and proprioceptive exercises on neck pain, neck function and neuropathic pain in patients with CR.

DETAILED DESCRIPTION:
Cervical radiculopathy is a common neck disorder that reduces function, productivity, and quality of life. Cervical radiculopathy impacts cervical nerves roots, with the highest prevalence of C6 and C7 nerve roots. The incidence of cervical radiculopathy affects roughly 107.3 out of 100,000 males and 63.5 out of 100, 000 females. This incidence in the fifth decade of life increases up to 203 per 100 000. The etiology of cervical radiculopathy is commonly attributed to mechanical compression or chemical irritation of the cervical nerve roots. The most contributing factor is probably related to disc herniation. Other problems that decrease the intervertebral foramen include trauma, infection, and tumors .

Inflammation or impingement of these nerve roots trigger pain receptors located in soft tissues and joints of the cervical spine, resulting in sensory changes such as tingling and motor loss in dermatomal and myotomal distribution depending on affected nerve root. Patients often complain of combination of neck pain and radiating pain in the arm. The impairments in cervical proprioceptive inputs have been attributed to neck pain and altered input from cervical afferents, particularly muscle spindle, Muscle spindles are accepted as being the primary cervical receptors responsible for position sense and are coupled to supplementary afferent input from the cutaneous and joint receptors.

Conservative treatment approaches described to date have included pharmacology, advice to remain active, manual therapy, exercise, acupuncture, traction, collars, epidural injection in addition to kinesio tape (KT). Manual therapy can include muscle energy techniques, high velocity manipulation or low velocity mobilization of the cervical and/or thoracic spine, soft-tissue mobilization, and neural mobilization techniques.

Previously, in different musculoskeletal problems, KT combined with conventional rehabilitation has been shown to produce greater improvements in pain, range of motion, and functional outcomes compared to the rehabilitation program alone in cervical spondylosis and low back pain. It was reported that in comparison to sham application, 2 weeks of kinesio tape (KT) application practiced in addition to a home exercise program was effective on pain and tenderness in individuals with cervical myofascial pain. Additionally, KT was effective on cervical proprioception 24 hours after its application in chronic neck pain patients. KT is believed to stimulate cutaneous and muscle mechanoreceptors, which enhances sensorimotor control and proprioceptive feedback, thereby assisting in movement coordination and reducing discomfort in ankle proprioception and different musculoskeletal conditions.

To date, there is only one study that specifically investigated the effect of KT on patient with CR. KT taping method along with manual therapy treatment, cervical stabilization exercises was effective in treating patients with cervical radiculopathy.

Exercise therapy is effective in the management of CR, which can relieve pain and improve cervical function. Many exercises used in management of CR like stretching exercises for tighten muscles. Neural mobilization techniques (e.g., Upper Limb Tension Test 1 sliding and gliding) to restore neural dynamics and decrease radicular pain .

Proprioceptive training can lead to significant improvements in proprioceptive and motor function across a range of healthy and clinical populations. General neck-shoulder ROM and cervical proprioceptive exercises including eye-head coordination exercise can be effective in improving neck proprioceptive acuity, pain, and disability in chronic nonspecific neck pain patients.

A study was conducted to investigate the effect of proprioceptive training on patients with CR, including cervical position sense training, head-eye coordination exercises, and postural control exercises. The authors reported a significant improvement in cervical ROM and marked reduction in pain intensity (VAS) in the proprioceptive training group compared to conventional physical therapy group.

The effectiveness of deep cervical flexors strengthening exercises has demonstrated positive outcomes in terms of decrease in neck pain and disability, improvement in sitting posture, enhanced neuromuscular control of the cervical flexors in patients with chronic neck pain, and improved proprioceptive acuity of the neck, indicating that proprioception can be enhanced with specific exercise.

Strengthening, stabilization, and eye-head coordination exercises directed toward the deep cervical flexors, scapular stabilizers, and oculomotor-cervical control has been shown to enhance cervical spine stability and improve proprioceptive function in neck pain.

To the best of the author's knowledge, no previous study combined proprioceptive exercises and Kinesio tape in management of CR. Consequently, this study will be conducted to examine the effect of this combination on proprioceptive in patients with CR.

ELIGIBILITY:
Inclusion Criteria:

* Age from 35-50years (Rafiq et al. 2022).
* BMI from 18 to 29.9 kg /m2 (Morsi et al., 2022.
* Current continuous or intermittent pain that has persisted for more than 3 months (Persson et al., 1997, Purves et al., 1998).
* Paresthesia or numbness along the course of the nerve (Young et al., 2009).
* Positive response for the 4 Wainner RS et al., test's item cluster:

  1. Ipsilateral cervical Spurling.
  2. Upper Limb Tension Tests (ULTTs).
  3. Neck Distraction.
  4. Spurling tests range (ROM) less than 60° (Wainner et al., 2003).
* Unilateral affection in the upper limb.

Exclusion Criteria:

* History of surgical procedures for pathologies giving rise to neck pain or CTS (Wainner et al., 2003).
* Clinical signs or symptoms of medical "red flags" or serious pathology (infection, cancer, and cardiac involvement) (George et al., 2015).
* Any systematic disease such as rheumatism and tuberculosis, cervical myelopathy, or multiple sclerosis (Joghataei et al., 2004).
* Systemic disease is known to cause generalized peripheral neuropathy as diabetes millitus (Wainner et al., 2003).
* Upper Motor neuron disease such as stroke and amyotrophic lateral sclerosis (ALS) (Joghataei et al., 2004).
* Complete loss of sensation along the involved nerve root (Moustafa & Diab, 2014).
* Primary report of bilateral radiating arm pain (Wainner et al., 2003)
* Pregnant woman (Moustafa & Diab, 2014).

Ages: 35 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Cervical proprioception | Baseline and 4 weeks
  The most common method used for assessment of cervical proprioception is Joint Position Error test, the active movement angle reproduction test, which requires the subject to relocate a neutral head position or a target head position selected by the investigator (Loudon et al., 1997; Hillier et al., 2015). In head position sense measurement studies, the variable measured is the difference between the reference point position entrenched initially (either a neutral or target position) and the position produced by the subject when attempting to match the target position , This difference is called JPE and has angular units of degrees (°) (Hillier et al., 2015). JPE test demonstrates good intra- and inter-rater reliability and acceptable validity for evaluating cervical proprioception (Revel et al., 1991; Kristjansson et al., 2003). JPE test will be measured by Laser Pointer Device.

SECONDARY OUTCOMES:
Cervical pain | at baseline and after 4 weeks
  The ANPRS is used to capture the patient's level of pain. It is an 11-point scale, ranging from 0 (no pain) to 10 (worst pain imaginable). The (NPRS) has been reported to be moderate (ICC value 0.63) in patients with CR (Cleland et al., 2006), and with acceptable reliability (ICC value 0.76) in patients with neck pain (Cleland et al., 2008).
Function | at baseline and after 4 weeks.
  The neck disability index (NDI) is the most widely used and validated instrument to assess the impact of neck pain on patients' functional activities and to measure outcomes in clinical practice and research. It consists of 10 questions: pain intensity, personal care, lifting, reading, headaches, concentration, work, driving, sleepi ng, and recreation (Vernon & Mior, 1991). The Arabic version of NDI is a condition-specific valid tool to assess the level of disabilities in patients with neck pain. The NDI-Ar is a reliable and valid questionnaire in neck pain patients with test-retest reliability; the ICC of the Arabic version was 0.96 (Shaheen et al., 2013).
Radicular pain | at baseline and after 4 weeks.
  The Upper Limb Tension Test 1 (ULTT1) will be used as both a screening tool for detecting radicular pain and as an outcome measure to evaluate changes in neural mobility and symptoms improvement throughout the intervention period.This test is commonly used in patients with cervical radiculopathy and has been shown to be both reliable and clinically relevant in identifying altered neural dynamics (Nee et al., 2012).

CONTACTS AND LOCATIONS:
Overall Officials: Eman A kamel, lecturer, Study Director — cairo university in Egypt

REFERENCES:
- [Result] Ferlinc A, Fabiani E, Velnar T, Gradisnik L. The Importance and Role of Proprioception in the Elderly: a Short Review. Mater Sociomed. 2019 Sep;31(3):219-221. doi: 10.5455/msm.2019.31.219-221. PMID 31762707
- [Result] Espi-Lopez GV, Aguilar-Rodriguez M, Zarzoso M, Serra-Ano P, Martinez DE LA Fuente JM, Ingles M, Marques-Sule E. Efficacy of a proprioceptive exercise program in patients with nonspecific neck pain: a randomized controlled trial. Eur J Phys Rehabil Med. 2021 Jun;57(3):397-405. doi: 10.23736/S1973-9087.20.06302-9. Epub 2020 Oct 13. PMID 33047944
- [Result] Caridi JM, Pumberger M, Hughes AP. Cervical radiculopathy: a review. HSS J. 2011 Oct;7(3):265-72. doi: 10.1007/s11420-011-9218-z. Epub 2011 Sep 9. PMID 23024624
- [Result] Agyenkwa SK, Mustafaoglu R, Yeldan I. Therapeutic Effects of Kinesiology Taping Versus Self-Mobilization on Neck Pain, Proprioception, Muscle Activity, and Respiratory Muscle Strength Among Prolonged Electronic Device Users. A Randomized Controlled Trial. Physiother Res Int. 2025 Apr;30(2):e70061. doi: 10.1002/pri.70061. PMID 40214192